CLINICAL TRIAL: NCT03615014
Title: Identification of Biopsychosocial Factors Predictive of the Post-traumatic Stress Disorder Occurrence in Patients Admitted to the Emergencies After Trauma
Brief Title: Predictive Factors of PTSD in Adults Admitted to an Emergency Service
Acronym: ISSUE
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Hospices Civils de Lyon (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: 69HCL18_0142
Record Dates: First submitted 2018-07-30; First posted 2018-08-03 (Actual); Last update posted 2025-12-19 (Actual); Status verified 2025-12

CONDITIONS: Post Traumatic Stress Disorder; Psychiatric Issue
MeSH Terms: conditions — Stress Disorders, Post-Traumatic

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Patients having trauma (Other): Adults patients having trauma in the month before visiting emergency will fill questionnaires
  Interventions: Other: Filling questionnaires

INTERVENTIONS:
Other: Filling questionnaires — Questionnaires will be submitted to patients during their visit to emergency service and 3 months later to evaluate the prevalence of Post Traumatic Stress Disorder and to identify predictive biopsychosocial factors

SUMMARY:
After trauma or stress factor like death exposition, serious injuries or sexual violence, some patients may develop stress reaction characterized by the presence of various symptoms among different categories (reviviscence, negative humor, dissociates symptoms, occasion, hypervigilance). In the month following trauma, the investigators speak of acute stress reaction (ASR) when symptoms are present during at least three days. If symptoms are present one month after trauma, then it is a post-traumatic stress disorder (PTSD).

Among patients visiting emergency after latest trauma, quite a few is in acute stress reaction. However, this reaction is often incorrectly identified by healthcare team, due to lack of oriented medical examination, patients visiting about other complaints (pain, insomnia) and not expressing clearly the trauma context. Yet, it is know that acute stress reaction occurrence and existence of dissociate symptoms after trauma confrontation is considerably predictive of the eventual post-traumatic stress disorder occurrence.

The identification of risk population of post-traumatic stress disorder is not the subject of any particular structured procedure in emergency services while early care of these patients may allow limiting post-traumatic stress disorder occurrence and associate consequences. Previous works on the subject having exclusively targeted some trauma subgroups or some predictive factors subtypes, investigators propose here biopsychosocial global approach that can weight the impact of each parameters.

In this study, investigators aim at determining predictive biopsychosocial factors of the post-traumatic stress disorder occurrence at 3 months in patients visiting emergency after latest trauma (less than one month old) and identified as "high-risk" to develop post-traumatic stress disorder (moderate or high).

ELIGIBILITY:
Inclusion Criteria:

* Man or woman aged between 18 and 70
* Admitted in an emergency service after a trauma less than one month old, defined by death exposition or death threat, serious injury or sexual violence, by one or several of the following;

  * Being directly exposed ;
  * Being direct witness of traumatic event that occurred to other people;
  * Hearing that traumatic event arrived to close family member or close friend. In the case of death penalty or death threat of a family member or a friend, events must have been violent or accidental.
  * Being exposed repeatedly or extremely to aversive characteristics of trauma events (for example: first line actors gathering human remains, cops exposed several times to kid sexual abuse explicit fact).
* Written informed-consent
* Affiliation to the French social security scheme or beneficiary of a similar scheme

Exclusion Criteria:

* Patient not understanding French language
* Patient under guardianship
* Clinical instability making impossible the realization of questionnaires (for example: agitation, vital risk, disorders of consciousness…)

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 460 (Actual)
Dates: Start 2019-02-11 (Actual); Primary Completion 2019-10-09 (Actual); Study Completion 2019-10-09 (Actual)

PRIMARY OUTCOMES:
Post Traumatic Stress Disorder (PTSD) occurrence | At 3 months following admission to the emergency service
  Presence or absence PTSD will be evaluated by the PCL-5 scale (PTSD Checklist for DSM-5 (Diagnostic and Statistical Manual of Mental Disorders -5)).
  The PCL-5 scale will be completed with patients during a phone interview with a psychologist or a psychiatrist.
  The PCL-5 is a 20-item questionnaire that assesses the 20 DSM-5 symptoms of PTSD.
  Patients will be asked to rate how bothered they have been by each item in the past 3-month on a 5-point Likert scale ranging from 0-4 (0 = not at all; 1 = a little bit; 2 = moderately; 3 = quite a bit; 4 = extremely).
  A provisional PTSD diagnosis can be made by treating each item rated as 2 = "Moderately" or higher as a symptom endorsed, then following the DSM-5 diagnostic rule which requires at least: 1 B item (questions 1-5), 1 C item (questions 6-7), 2 D items (questions 8-14), 2 E items (questions 15-20).
  Items are summed to provide a total score. The range is 0-80. A total score of 33 or higher signifies the likely presence of PTSD.

SECONDARY OUTCOMES:
Prevalence of high risk patients to develop Post Traumatic Stress Disorder | 1 day (at admission to the emergency service)
  The high risk of developing Post Traumatic Stress Disorder will be determined by the Impact of Event Scale-Revised (IES-R).
  The IES-R is a 22-item self-report questionnaire that assesses subjective distress caused by traumatic events. The IES-R contains sub-scales for avoidance, intrusions and hyperarousal.
  Patients will be asked to indicate how much they were distressed or bothered during the past seven days by each item.
  Items are rated on a 5-point scale ranging from 0-4 (0 = not at all; 1 = a little bit; 2 = moderately; 3 = quite a bit; 4 = extremely). The IES-R yields a total score ranging from 0 to 88.
  A total IES-R score of over 34 signifies patient is at high risk to develop PTSD.
Prevalence of moderate risk patients to develop Post Traumatic Stress Disorder | 1 day (at admission to the emergency service)
  The moderate risk of developing Post Traumatic Stress Disorder will be determined by the Impact of Event Scale-Revised (IES-R).
  The IES-R is a 22-item self-report questionnaire that assesses subjective distress caused by traumatic events. The IES-R contains sub-scales for avoidance, intrusions and hyperarousal.
  Patients will be asked to indicate how much they were distressed or bothered during the past seven days by each item.
  Items are rated on a 5-point scale ranging from 0-4 (0 = not at all; 1 = a little bit; 2 = moderately; 3 = quite a bit; 4 = extremely). The IES-R yields a total score ranging from 0 to 88.
  An IES-R score between 12 and 34 included signifies patient is at moderate risk to develop PTSD.
Post Traumatic Stress Disorder incidence | At 3 months following admission to the emergency service
  Presence of Post Traumatic Stress Disorder will be determined by the PCL-5 scale at 3 months following admission to the emergency service (primary outcome measure). Incidence is the rate of newly diagnosed patients of PTSD at 3 months.
Dissociative experiences | At admission to the emergency service
  Describe the patient dissociative disorders using the Questionnaire of Peritraumatic Dissociative Experiments score.
  The Peritraumatic Dissociative Experiences Questionnaire (PDEQ) determines the presence and the intensity of the peritraumatic response experienced by the individual at the time of the traumatic event, and in the minutes and hours that followed.
  The PDEQ in a 10-item test. Each item is scored from 1 (not at all true) to 5 (extremely true). The total score is the sum of all items. A score above 15 is indicative of significant dissociation.
Social consequences | At 3 months following admission to the emergency service
  Describe Post Traumatic Stress Disorder impact on social life using the Social Support Questionnaire (SSQ6).
  The Social Support Questionnaire 6 (SSQ6) is a 6-item questionnaire designed to measure two dimensions of social support: availability and satisfaction.
  Each item is a question that solicits a two-part answer: Part 1 asks participants to list up nine people maximum available to provide support in each of 6 areas, and Part 2 asks participants to indicate how satisfied they are, in general, with these people.
  Availability is scored by counting the total number of people for each item (max = 54), and satisfaction is scored by counting the total satisfaction scores for the 6 items (max = 36).
Social consequences | At 3 months following admission to the emergency service
  Describe PTSD impact on professional life by calculating the number of sick leave days over the 3 months
Complications associated to Post Traumatic Stress Disorder | At 3 months following admission to the emergency service
  Impact of the excessive drinking and alcohol using the Alcohol Use Disorders Identification Test (AUDIT) at 3 months.
  The AUDIT is a 10-item screening tool that assesses alcohol consumption, drinking behaviors, and alcohol-related problems. Each item has a score ranging from 0 to 4.
  Total scores of 7 or more in men, 6 or more in women are recommended as indicators of hazardous and harmful alcohol use.
Complications associated to Post Traumatic Stress Disorder | At 3 months following admission to the emergency service
  Impact of the nicotine dependence at 3 months using the Fagerström test. The Fagerström Test is a standard instrument for assessing the intensity of physical addiction to nicotine.
  In scoring the Fagerstrom Test, yes/no items are scored from 0 to 1 and multiple-choice items are scored from 0 to 3. The items are summed to yield a total score of 0-10.
  A patient who scores between 0 and 2 is classified as no nicotine dependence; a score of 3 or 4 would be considered to have low dependence on nicotine, moderate dependence for a score of 5 or 6, high dependence for a score of 7 or 8, and very high dependence for a score of 8 or over.
Complications associated to Post Traumatic Stress Disorder | At 3 months following admission to the emergency service
  The severity of depressive symptoms at 3 months will be determined by the 16-item Quick Inventory of Depressive Symptomatology (QIDS-SR16).
  The QIDS-SR 16 is a self-report questionnaire that assesses the severity of depressive symptoms. The 16 items (questions) on the QIDS-SR16 cover the nine diagnostic symptom criteria used in DSM.
  Each item is rated 0-3. The QIDS-SR16 is scored by summing responses for each of the 16 items to obtain a total score ranging from 0 to 27.
  A total score from 0 to 5 signifies absence of depression; 6 to 10 mild depression; 11 to 15 moderate depressions, 16 to 20 severe depression and from 21 to 27 very severe depression.

CONTACTS AND LOCATIONS:
Overall Officials: Clémence BIED, Dr, Principal Investigator — Hospices Civils de Lyon
Locations (5):
- France (5):
  - CHU Clermont - Hôpital G Montpied - Urgences Psychiatriques et Médecine d'urgence, Clermont-Ferrand
  - CH St Joseph St Luc - Urgences Psychiatriques et Médecine d'urgence, Lyon
  - Hôpital Edouard Herriot - Urgences Psychiatrique et Médecine d'urgence, Lyon
  - Centre Hospitalier Lyon Sud - Urgences psychiatriques, Pierre-Bénite
  - CHU St Etienne - Hôpital Nord - Urgences Psychiatriques, Saint-Priest-en-Jarez

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Wafa MH, Viprey M, Magaud L, Haesebaert J, Leaune E, Poulet E, Bied C, Schott AM. Identification of biopSychoSocial factors predictive of post-traUmatic stress disorder in patients admitted to the Emergency department after a trauma (ISSUE): protocol for a multicenter prospective study. BMC Psychiatry. 2019 May 30;19(1):163. doi: 10.1186/s12888-019-2154-z. PMID 31146712